CLINICAL TRIAL: NCT03225053
Title: EFFECTS OF MIOFASCIAL RELEASE AND PERCUTANEOUS MICROELETROLYSIS IN INDIVIDUALS WITH TYPICAL TYPE HEADACHE
Brief Title: EFFECTS OF MIOFASCIAL RELEASE AND PERCUTANEOUS MICROELETROLYSIS IN TYPE HEADACHE
Acronym: EMRPMITH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rodrigo Marcel Valentim da Silva (Other)
Responsible Party: Sponsor-Investigator, Rodrigo Marcel Valentim da Silva, Principal Investigator, Estácio Ponta Negra
Organization: Estácio Ponta Negra (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RSilva
Record Dates: First submitted 2017-06-11; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Trigger Point; Tension-Type Headache
Keywords: Percutaneous microelectrolysis; Physiotherapy
MeSH Terms: conditions — Tension-Type Headache | interventions — Heart Rate

STUDY DESIGN:
Intervention Model Description: After the initial evaluation, the investigator 2 will conduct the experimental procedures in the different groups, which will be submitted to the following protocols: G1 (n = 15) called LMF will be submitted to the myofascial release technique consisting of: , Deep sliding, pumping-kneading, thumb and four-finger rubbing, and sliding) applied to the musculature of the most painful region for 15 minutes. G2 (n = 15) will be applied to the MEP® technique, in which needles will be introduced on three occasions during each session, at different points of the musculature of the most painful region, for a total of 3 minutes. The G3 (n = 15) will be performed the two techniques above, being applied first Miofascial Release and later to MEP®. G4 (n = 15) will be the control group, not performing any of the interventions. The reevaluations will occur immediately and after 48 hours of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MEP® technique (Experimental): G1 (n = 15), referred to as LMF, will be submitted to the myofascial release technique consisting of: classic massage (superficial sliding, deep sliding, pumping-kneading, pulse and four-finger smear and sliding) Minutes. G2 (n = 15) will be applied to the MEP® technique, in which the needles will be introduced in three occasions during each session, in different points of the musculature of the most painful region, for a total of 3 minutes. The G3 (n = 15) will execute the two techniques above, being applied the first version Myofascial and later to the MEP®. G4 (n = 15) will be the control group, not performing any of the interventions. The reevaluations will occur immediately and after 48 hours of the intervention.
  Interventions: Device: MEP® technique

INTERVENTIONS:
Device: MEP® technique — G1 (n = 15), referred to as LMF, will be submitted to the myofascial release technique consisting of: classic massage (superficial sliding, deep sliding, pumping-kneading, pulse and four-finger smear and sliding) Minutes. G2 (n = 15) will be applied to the MEP® technique, in which the needles will be introduced in three occasions during each session, in different points of the musculature of the most painful region, for a total of 3 minutes. The G3 (n = 15) will execute the two techniques above, being applied the first version Myofascial and later to the MEP®. G4 (n = 15) will be the control group, not performing any of the interventions. The reevaluations will occur immediately and after 48 hours of the intervention.
  Other Names: classic massage (superficial sliding, deep sliding, pumping-kneading, pulse and four-finger smear and sliding)

SUMMARY:
A headache is a more common disorder and one that prevails over a lifetime of much of the population. Among the causes are in the stress and spasms of the pericranial musculature, presence of painful sensitivity in the region, decrease of pain threshold, and a presence of trigger points (PGs) that can also cause as headaches. The solutions for health and health, in addition to Percutaneous Microelectrolysis (MEP®), which is used in the application of low intensity galvanic current through the acupuncture needle. Although it is a very common pathology, it is still little studied and a lack of information is a question of solutions such as crisis of care. This work justifies the negative bones of CTT in university students, as this has repercussions on the quality of life, besides proposing a therapeutic approach to reduce the symptomatology. The present study aims to investigate the effects of myofascial release techniques, MEP® and an association of therapies, observing the impact on quality of life and repercussions on academic performance. This is a controlled clinical trial of a convenience-based approach, consisting of universities between the 1st and 10th Physical Therapy course of Estácio Ponta Negra, over 18 years of age, who are not present in the application of the questionnaires, It is necessary to use the medicine of the analgesic type. The volunteers are evaluated through the HIT-6 and SF-36 questionnaires, after a selection of pain evaluation, PGs and algometry. The randomization will consist of 4 groups, after a consultation and an immediate re-evaluation and a second time and a new intervention and re-evaluation. A descriptive and inferential statistics will be performed through the SPSS 20.0 program. The normality of the data is observed by the Kolmogorov-Smirnov (KS) test. For a comparison between groups whose parametric data are applied or anova test with post hoc tukey comingue of significance of 5% (p <0.05). It is believed that the use of the association of myofascial release techniques and Percutaneous Microelectronics promotes greater benefits in tension headache.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old, they will be present at the time of ordering, not being pregnant and not taking analgesic medication at least 24 hours before the intervention.

Exclusion Criteria:

* More than 20% of the questionnaire data are incomplete and if during the research the volunteer presents some discomfort.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-20 (Estimated); Primary Completion 2017-12-20 (Estimated); Study Completion 2018-01-30 (Estimated)

PRIMARY OUTCOMES:
Headache impact test (HIT-6) | ten minutes
  This is composed of six questions, with scores ranging from six to 13 points, which can total between 36-78 points; So the higher this score, the greater the impact of headache on the daily activities of the individual.
Quality of life assessment (SF-36) | ten minutes
  Validated and adapted to the Brazilian culture. This allows to compare the quality of life of healthy individuals and patients of different pathologies. It consists of 36 questions, which encompass 8 components: functional capacity, physical aspects, pain, general health, vitality, social aspects, emotional aspects and mental health. The final score can vary from 0 (worst general health condition) to 100 (better health).
Pain assessment | five minutes
  To grade the pain before the intervention will be applied the visual analogue scale. It is a subjective test in which the volunteer will self-evaluate. It will be performed with a horizontal line in which the beginning will represent absence of pain and at the end of the line will represent the maximum pain, and will be oriented to mark in the line the perception of the pain at that moment.
Evaluation of trigger points | twenty minutes
  The presence of trigger points in the upper trapezius, sternocleidomastoid, suboccipital and splenius muscles of the neck will be investigated. Localization along the tense muscle band to the presence of palpable nodules, local pain to the digital compression (estimated time of 6 s) of a palpable nodule located in a tight band; Recognition of pain referred by the patient as familiar by pressing the sensitive nodule (to identify active PG)
Assessment of pressure pain threshold | twenty minutes
  To evaluate the pain threshold, a WAGNER FDX algometer will be used, which is a device consisting of a rubber disk measuring 1 cm2 connected to a pressure gauge, which has values in kgf / cm2. The upper trapezius muscle will be evaluated at the mean distance between the C7 and the acromion of the scapula along its fibers. If the algometry evaluation point coincides with the trigger point, the analysis with the algometer will be performed 2 cm apart in the medial to the point direction.

IPD SHARING:
Plan to Share IPD: No